CLINICAL TRIAL: NCT01681719
Title: Whole Body Vibration as Alternative for Improve the Ergospirometric Values in Elderly: a Randomized Clinical Trial
Brief Title: Ergospirometric Values and WBV in Elderly
Acronym: EVAWIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Principal Investigator, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ERGOFORCE1
Record Dates: First submitted 2012-08-30; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Aging
Keywords: VO2; VCO2; VE/VO2; heart rate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WBV and resistance (Experimental): used both interventions
  Interventions: Device: WBV and Resistance
- WBV & resistance sham (Experimental): used the vibrating platform and sham for resistance training
  Interventions: Device: WBV & resistance sham
- Resistance & sham WBV (Experimental): used resistance exercises and sham for vibrating platform
  Interventions: Device: resistance & sham WBV

INTERVENTIONS:
Device: WBV and Resistance — use of WBV and resistance device during 03 months in elderly health people. The WBV used progressive increases of time and amplitude and the resistance training improves the weight.
  For Resistance: performed in upper and lower limbs in weight machine Mega II Movement®, used guidelines from American College of Sports Medicine for elderly, with two series of 08 repetitions (75% weight of one RM), considered for RM calculation the maximum voluntary isometric contraction.
  For WBV: used MY3 platform (Power Plate®, MY3, UK) frequency 35 hertz, tri-axial, amplitude 02 mm in adaptation and initial phases, increasing to 04 mm in phases intermediate and final. The time initial was 10 minutes, progressed to 15 min in second month, concluding with 20 min. Rest time between series remained 01 min.
  Arms: WBV and resistance
Device: resistance & sham WBV — used only resistance
  For Resistance: performed in upper and lower limbs in weight machine Mega II Movement®, used guidelines from American College of Sports Medicine for elderly, with two series of 08 repetitions (75% weight of one RM), considered for RM calculation the maximum voluntary isometric contraction.
  For WBV: used MY3 platform (Power Plate®, MY3, UK)off.
  Arms: Resistance & sham WBV
Device: WBV & resistance sham — used really the WBV, but sham for resistance training
  For Resistance: performed similar movments in upper and lower limbs in weight machine Mega II Movement®, without using weights.
  For WBV: used MY3 platform (Power Plate®, MY3, UK) frequency 35 hertz, tri-axial, amplitude 02 mm in adaptation and initial phases, increasing to 04 mm in phases intermediate and final. The time initial was 10 minutes, progressed to 15 min in second month, concluding with 20 min. Rest time between series remained 01 min.
  Arms: WBV & resistance sham

SUMMARY:
this study aims evaluate the ergospirometric values after 03 months of training with WBV in elderly health people. The hypothesis is increases of ergospirometric values.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-74 years,
* Sedentary or Moderate A in accord with IPAQ short form (International Physical Activity Questionnaire) and those without disease.
* furthermore, the subjects should reach the ventilatory threshold 1, considered after meeting two of the following events:
* respiratory quotient (R) increases (R ≥1,1);
* loss of linearity between the pulmonary ventilation curve (VE) and oxygen consumption (VO2), plateau of VO2 or plateau of heart rate (HR) and increases of end-tidal PO2 (Pet O2)

Exclusion Criteria:

* Were excluded subjects with changes in Mini-mental state examination (MMSE) scores by age and educational level where the minimum score represents: illiterate 13 points, less than 8 study years is 18 points, 8 or more study years is 26 points 11.
* Were also excluded current smokers or previous, subjects with thrombosis, labyrinthitis, diabetes, hemodynamic instabilities, obesity, osteoporosis, neuromuscular diseases, pulmonary or cardiac diseases, changes in resting electrocardiogram or in exercise, ingestion of drugs to metabolism bone / muscle / heart chronotropism or with difficulties in adapting protocols

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
maximal O2 consumption | started and finished the protocol after 03 months

CONTACTS AND LOCATIONS:
Locations (1):
- UFPE, Recife, Pernambuco, Brazil